CLINICAL TRIAL: NCT07345910
Title: Decoding the Triad: the Interplay Between Environment, Pathogen, and Host in Melioidosis (DeEPH)
Brief Title: Environment, Pathogens, and Host Interactions in Melioidosis
Acronym: DeEPH
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: MEL25001
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Melioidosis
MeSH Terms: conditions — Melioidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for the following analyses:
  * DNA for genetic profiling
  * Serum for antibody measurement
  * Peripheral blood mononuclear cells (PBMCs) for immune cell analysis
  * HbA1c for assessment of blood glucose control
  * Plasma lactate for marker for disease severity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Melioidosis patients: Patients confirmed to have melioidosis
- Healthy controls: Healthy controls will be enrolled for each confirmed melioidosis case. A healthy control is defined as an individual with no current fever, no evidence of soft tissue infection, and no prior history of melioidosis. Controls will be recruited within approximately two weeks of case identification and will be matched to cases by age (±5 years), sex, and village of residence.
- Sandbox village cohort: All residents of the Sandbox Village, a high-risk area for melioidosis, will be enrolled to monitor disease progression and to evaluate the impact of improved water sanitation.

SUMMARY:
This is a longitudinal, multicentre observational study conducted across three established microbiology units integrated within hospital and community health systems in Thailand, Lao PDR, and Cambodia.

The hospital cohort will enroll approximately1,000 patients with positive melioidosis. Participants will be followed at six time points from admission through one year (post-discharge) to capture acute and recovery-phase outcomes, with clinical data collected on demographics, comorbidities, exposures, treatment, adherence, and outcomes.

For each confirmed case, a healthy control will be recruited within two weeks and matched by age, sex, and village of residence. Controls with no symptoms or history of melioidosis will provide a single blood sample at enrolment and will be followed by telephone at 6 and 12 months.

In addition to hospital-based surveillance, a high-risk community in northern Ubon Ratchathani-referred to as the Sandbox Village-will be intensively monitored to capture subclinical infections and to assess environmental factors influencing disease acquisition.

This study is funded by the Wellcome Trust. The grant reference number is 323077/Z/24/Z

DETAILED DESCRIPTION:
This is a longitudinal, multicentre observational study conducted across three established microbiology units integrated within hospital and community health systems:

* Sunpasitthiprasong Hospital, Ubon Ratchathani, Thailand (MORU);
* Mahosot Hospital, Vientiane, Lao PDR (LOMWRU); and
* Angkor Hospital for Children, Siem Reap, Cambodia (COMRU).

In addition to hospital-based surveillance, a high-risk community in northern Ubon Ratchathani-referred to as the Sandbox Village-will be intensively monitored to capture subclinical infections and to assess environmental factors influencing disease acquisition.

Participant Recruitment and Follow-up

Hospital cohort:

Patients with melioidosis will be recruited at all three hospital sites. The study plans to recruit 1,000 patients, who will be followed longitudinally at six time points: Day 0 (admission), Days 3 and 7 (acute phase), and Days 30, 180, and 365 (recovery phase).

Clinical data collected will include demographic characteristics, underlying comorbidities, environmental exposures, lifestyle and behavioural factors, treatment history, patient-reported medication adherence, and follow-up outcomes.

Healthy controls:

Each patient will be matched with a healthy control recruited within two weeks of diagnosis, based on age, sex, and village of residence. Controls will have no current symptoms or prior history of melioidosis. They will provide a single blood sample at enrolment for DNA extraction and antibody profiling and will be followed up by telephone on Days 180 and 365.

Community cohort:

To complement hospital-based data and to identify subclinical infections, intensive community surveillance will be conducted in the Sandbox Village, a high-incidence area within the Ubon Ratchathani region. All residents (approximately 400 individuals) will be enrolled. DNA samples will be collected at baseline, and serum samples will be obtained every two months over a 42-month period, either at participants' homes or at a central village location, to measure antibody responses to Burkholderia pseudomallei as a proxy for exposure.

Community cohort:

To complement hospital-based data and to identify subclinical infections, intensive community surveillance will be conducted in the Sandbox Village, a high-incidence area within the Ubon Ratchathani region. All residents (approximately 400 individuals) will be enrolled. DNA samples will be collected at baseline, and serum samples will be obtained every two months over a 42-month period, either at participants' homes or at a central village location, to measure antibody responses to Burkholderia pseudomallei as a proxy for exposure.

ELIGIBILITY:
Inclusion criteria for melioidosis patients:

* Age ≥20 years
* Positive for Burkholderia pseudomallei from any clinical samples
* Resident of the study area for at least two years, including the follow-up period
* Willing to participate and give informed consent.

Inclusion criteria for healthy controls:

* Age ≥20 years
* Currently healthy as judged by study doctor
* Resident of the study area for at least two years, including the follow-up period
* Willing to participate and give informed consent.

Inclusion criteria for sandbox residents:

* Age ≥20 years
* Resident of the study area for at least two years, including the follow-up period
* Willing to participate and give informed consent.

Exclusion criteria for melioidosis patients:

* Current tuberculosis (TB) or TB treatment within the past six months
* Documented HIV infection or use of immunosuppressive therapy in the past 12 months

Exclusion criteria for healthy controls:

* History of melioidosis
* Significant acute illness
* Current fever or soft tissue infection

Exclusion criteria for sandbox residents

-N/A

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Melioidosis patients:
  Patients confirmed to have melioidosis.
  Healthy controls:
  For each confirmed melioidosis case, a healthy control-defined as having no current fever, no evidence of soft tissue infection, and no prior history of melioidosis-will be recruited from satellite blood bank donors within approximately two weeks of case identification. Controls will be matched by age (±5 years), sex, and village of residence.
  Sandbox Village residents:
  All residents of the Sandbox Village, a high-risk area for melioidosis, will be enrolled to monitor disease progression and to evaluate the impact of improved water sanitation.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2034-12-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Development of melioidosis following exposure, assessed among melioidosis cases | 365 days
Development of melioidosis following exposure, assessed among healthy controls | 365 days
Development of melioidosis following exposure, assessed among Sandbox Village residents | 3.5 years
Mortality during the acute phase of infection among individuals with melioidosis (melioidosis cases). | 365 days
Number of hospital readmissions following discharge among individuals with melioidosis (melioidosis cases). | 365 days

SECONDARY OUTCOMES:
Changes in disease development following exposure associated with interactions between environmental modifications. | 3.5 years
Changes in mortality during the acute phase of infection following exposure associated with interactions between environmental modifications. | 365 days
Changes in hospital readmission following recovery associated with interactions between environmental modifications. | 365 days
Changes in disease development following exposure associated with interactions between clinical management factors. | 365 days
Changes in mortality during the acute phase of infection following exposure associated with interactions between clinical management factors. | 365 days
Changes in hospital readmission following recovery associated with interactions between clinical management factors. | 365 days
Changes in disease development following exposure associated with interactions involving genetic susceptibility. | 365 days
Changes in mortality during the acute phase of infection following exposure associated with interactions involving genetic susceptibility. | 365 days
Changes in hospital readmission following recovery associated with interactions involving genetic susceptibility. | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Kamolchanok Claire Chewapreecha, PhD, Principal Investigator — Mahidol Oxford Tropical Research Unit
Locations (3):
- Cambodia-Oxford Medical Research Unit (COMRU), Siem Reap, Cambodia
- Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (LOMWRU), Vientiane, Laos
- Sunpasitthiprosong Hospital, Ubon Ratchathani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The study outputs, including genomic and transcriptomic data and associated metadata, will be valuable for future research. In compliance with the Wellcome Trust's open data policies and to encourage reproducibility, data will be deposited in two repositories:
  Human genomic and transcriptomic data: European Genome-Phenome Archive (EGA), under managed access
  Bacterial genomic data: European Nucleotide Archive (ENA), open access
  Pseudonymised metadata, including participant demographics and microbiological findings, will be shared with qualified researchers in accordance with the General Data Protection Regulation (GDPR). No personally identifiable information will be shared, and participants will not be identifiable from any released data.
Supporting Information: Study Protocol